CLINICAL TRIAL: NCT02531399
Title: Measurement of Total Retinal Blood Flow During Flicker Stimulation in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-250315
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: flicker induced changes; total volumetric retinal blood flow
MeSH Terms: interventions — Laser-Doppler Flowmetry

ARMS (1):
- Healthy Subjects (Experimental): 20 healthy female and male volunteers, age 18-45 years, non-smokers. Measurements with FDOCT, DVA, LDV and LSFG will be done in all healthy subjects.
  Interventions: Device: FDOCT; Device: LDV; Device: DVA; Device: LSFG

INTERVENTIONS:
Device: FDOCT — Measurement of retinal blood velocities
  Other Names: Fourier Domain Color Doppler Optical Coherence Tomography
Device: LDV — Measurement of retinal blood velocities
  Other Names: Laser Doppler Velocimetry
Device: DVA — Measurement of retinal vessel diameters
  Other Names: Dynamic Vessel Analyzer
Device: LSFG — Imaging of retinal blood flow
  Other Names: Laser Speckle Flowgraphy

SUMMARY:
Neurovascular coupling or functional hyperemia is defined as an essential physiologic mechanism in the brain, which is necessary for the local adaption of blood flow to altered metabolic demands of the tissue. It has been shown that also in the eye, blood flow is considerably coupled to retinal neural activity. The current concept of functional hyperemia is that visual stimulation, as flicker light, effectuates increasing neural activity in the retina, which elevates the metabolic needs of the retinal tissue for oxygen and glucose and consequently induces dilatation and augmented blood flow in the retinal vasculature. In several studies, stimulation with flicker light has been shown to induce an increase of blood flow in major retinal arteries and veins as well as an increase of optic nerve head blood flow. Up until now, flicker induced changes in blood flow were measured solely in the major retinal arteries and veins with systems such as the commercially available dynamic vessel analyzer (DVA) by Imedos and with laser Doppler velocimetry (LDV).

In the present study, the investigators propose to measure the response of total retinal blood flow to diffuse luminance flicker stimulation with bi-directional Fourier Domain Doppler Optical Coherence Tomography (FDOCT) as well as with Laser Speckle Flowgraphy (LSFG) in healthy subjects by assessing vessel diameter, blood velocity and blood flow of all retinal vessels. For comparative reasons, the investigators will furthermore assess the blood flow of major retinal arteries and veins with the dynamic vessel analyzer (DVA) and laser Doppler velocimetry (LDV).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent for participation
* Men and women aged between 18 and 45 years
* Non-smokers
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Systolic blood pressure < 140 mmHg, diastolic blood pressure < 90 mmHg
* Normal ophthalmic findings, ametropia less than 3 diopters

Exclusion Criteria:

* History or presence of ocular disease
* Ametropy ≥ 3 dpt
* Treatment with any drug in the 3 weeks preceding the first study day
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Participation in a clinical trial in the 3 weeks preceding the first study day
* Blood donation during the 3 weeks preceding the first study day
* History of family history of epilepsy
* Abuse of alcoholic beverages
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Flicker induced changes in total retinal blood flow (FDOCT) | 1 day

SECONDARY OUTCOMES:
Red blood cell velocity (LDV) | 1 day
Retinal vessel diameters (DVA) | 1 day
Retinal oxygen saturation (DVA) | 1 day
Relative Flow Volume (LSFG) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhoefer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Austria, Vienna, Austria

REFERENCES:
- [Derived] Fondi K, Aschinger GC, Bata AM, Wozniak PA, Liao L, Seidel G, Doblhoff-Dier V, Schmidl D, Garhofer G, Werkmeister RM, Schmetterer L. Measurement of Retinal Vascular Caliber From Optical Coherence Tomography Phase Images. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT121-9. doi: 10.1167/iovs.15-18476. PMID 27409462